CLINICAL TRIAL: NCT07277816
Title: Photo-experiencing and Reflective Listening (PEARL) to Promote Healing Engagement for Survivors of Violence: A Feasibility Study
Brief Title: Photo-experiencing and Reflective Listening (PEARL) to Promote Healing Engagement for Survivors of Violence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 272926; 5K01NR021275-02 (NIH)
Record Dates: First submitted 2025-12-01; First posted 2025-12-11 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Violence and Victimization
Keywords: healing; recovery; violence; trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participants are randomized to receive the PEARL intervention either immediately or after a 3-month waiting period, with the waitlist control group crossing over to receive the intervention after their waiting period ends.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Experimental): Participants randomized to this arm receive the PEARL intervention within two weeks of enrollment. They are given a photography-focusing prompt and two weeks to create photographs reflecting their healing journey. After two weeks, they participate in a reflective listening interview about their photographs. Participants complete surveys at baseline, immediately post-intervention, and at one-month follow-up, as well as a qualitative interview at one-month follow-up.
  Interventions: Behavioral: PEARL (Photo-experiencing and Reflective Listening)
- Waitlist Control Group (Active Comparator): Participants randomized to this arm receive a resource referral list (standard of care) and wait three months before receiving the PEARL intervention. They complete baseline surveys at enrollment and again at three months (pre-intervention baseline). After the three-month waiting period, they receive the same PEARL intervention as the immediate group: a photography-focusing prompt, two weeks to create photographs, and a reflective listening interview. They complete post-intervention and one-month follow-up assessments following their intervention.
  Interventions: Behavioral: PEARL (Photo-experiencing and Reflective Listening)

INTERVENTIONS:
Behavioral: PEARL (Photo-experiencing and Reflective Listening) — PEARL is a two-component behavioral intervention designed to promote healing engagement among survivors of interpersonal violence. Participants receive a photography-focusing prompt and are given two weeks to create photographs that reflect their healing journey and experiences. After the two-week photography period, participants engage in a one-on-one reflective listening interview where they discuss the photographs they created and co-create a healing action plan based on these discussions. The interview provides a structured opportunity for participants to explore and articulate their healing process through photo-elicitation, allowing them to express their experiences visually and verbally. The intervention is delivered by trained research assistants with fidelity monitoring through audio recording and independent evaluation of a random sample of sessions.
  Other Names: Photo-elicitation intervention for trauma survivors

SUMMARY:
The goal of this clinical trial is to learn if a photo-elicitation intervention called PEARL (Photo-experiencing and Reflective Listening) can promote healing engagement in survivors of interpersonal violence. It will also learn about the feasibility and acceptability of PEARL. The main questions it aims to answer are:

Does PEARL reduce barriers to help-seeking for trauma? Does PEARL improve trauma coping self-efficacy? Does PEARL change post-trauma cognitions and readiness for recovery? Is PEARL feasible and acceptable to survivors of interpersonal violence?

Researchers will compare people who receive PEARL immediately to people on a waitlist (who receive PEARL three months later) to see if PEARL improves healing engagement and help-seeking behaviors.

Participants will:

* Complete baseline surveys about their trauma history, mental health, healing, and help-seeking behaviors
* Be randomly assigned to receive PEARL immediately or after a 3-month wait
* Receive a photography-focusing prompt and create photos over two weeks (those in the immediate group or after the waiting period)
* Participate in a reflective listening interview about their photos
* Complete follow-up surveys immediately after the intervention and one month later
* Participate in a one-month follow-up interview about their experience

DETAILED DESCRIPTION:
This is a randomized waitlist control feasibility study of the PEARL (Photo-experiencing and Reflective Listening) intervention for women survivors of interpersonal violence. The study will enroll 40 participants recruited through local community organizations, interpersonal violence email listservs, and social media platforms.

Randomization and Study Arms:

Interested participants will complete an online baseline questionnaire through Qualtrics and be randomly assigned (1:1) to either:

1. Immediate Intervention Group (n=20): Receives PEARL within two weeks of enrollment
2. Waitlist Control Group (n=20): Receives a resource referral list (standard of care) and completes PEARL three months later

Intervention Protocol:

The PEARL intervention consists of two components:

1. Participants receive a photography-focusing prompt and have two weeks to create photographs
2. Participants complete a reflective listening interview about their photographs

Assessment Schedule:

* Baseline: Demographics, trauma history, and outcome measures
* Post-intervention: Outcome measures completed immediately after the intervention (trauma coping self-efficacy, post trauma cognitions, healing)
* One-month follow-up: Outcome measures and qualitative interview (trauma coping self-efficacy, post trauma cognitions, healing, help-seeking actions, depression, anxiety, PTSD).

The waitlist control group completes an additional baseline survey three months after initial enrollment, which serves as their pre-intervention assessment.

Data Analysis: Feasibility will be assessed through completion rates, and research assistant evaluations. Acceptability will be evaluated through participant surveys and follow-up interviews. Preliminary impact on healing engagement and help-seeking will be analyzed using descriptive statistics and nonparametric tests. Qualitative data from open-ended survey questions, research assistant evaluations, and follow-up interviews will undergo thematic analysis. Quantitative and qualitative findings will be integrated to provide a comprehensive understanding of PEARL's feasibility, acceptability, and potential impact.

Community Engagement: The study incorporates feedback from Community Advisory Board (CAB) and Scientific Advisory Board (SAB) members throughout the research process. Purposive sampling strategies will be employed to achieve maximum diversity in participant age.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* History of interpersonal violence (IV) - identifies as a survivor of interpersonal violence
* Able to complete an interview in English
* Able to provide informed consent

Exclusion Criteria:

* Under 18 years of age
* Does not identify as a woman (male participants excluded)
* No history of interpersonal violence
* Unable to complete an interview in English
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Post-trauma Cognitions Inventory (PTCI) | Baseline, immediately post-intervention (approximately 2-4 weeks after baseline), and 1-month follow-up (approximately 6-8 weeks after baseline)
  The PTCI is a self-report measure used to assess posttraumatic cognitions. It is composed of three subscales: Negative Cognitions about the Self, Negative Cognitions about the World, and Self-Blame. Higher scores indicate more negative trauma-related cognitions. The minimum score one can receive is 33 and the maximum score is 231.
Trauma Coping Self-efficacy Scale | Baseline, immediately post-intervention (approximately 2-4 weeks after baseline), and 1-month follow-up (approximately 6-8 weeks after baseline)
  The Trauma Coping Self-efficacy Scale is a 7-item measure that covers trauma-related coping self-efficacy including: dealing with reminders of the event, dealing with emotions associated with the event, employing active coping strategies, and resuming normal functioning. Higher scores indicate greater confidence in ability to cope with trauma. The minimum score one can receive is 0 and the maximum score is 63.
Healing after Gender-based Violence Scale | Baseline, immediately post-intervention (approximately 2-4 weeks after baseline), and 1-month follow-up (approximately 6-8 weeks after baseline)
  This 18-item scale measures holistic healing after trauma. Items are rated on a 5-point Likert scale from 1 ('Not at all') to 5 ('To a great extent'). Respondents are asked to evaluate each statement in reference to their perceived lowest point and their current feelings. This measure captures holistic healing outcomes beyond symptom reduction. Higher scores indicate greater levels of healing.

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Baseline and 1-month follow-up (approximately 6-8 weeks after baseline)
  The PCL-5 is a 20-item self-report measure that assesses the presence and severity of PTSD symptoms according to DSM-5 criteria. Response options are on a 5-point Likert scale with anchors: 0 = not at all, 4 = extremely. Items assess intrusion symptoms, avoidance, negative alterations in cognitions and mood, and alterations in arousal and reactivity. A total symptom severity score (range 0-80) can be obtained by summing the scores for each of the 20 items. A score of 33 is the current clinical cut-off for probable PTSD.
Patient Health Questionnaire-8 (PHQ-8) | Baseline and 1-month follow-up (approximately 6-8 weeks after baseline)
  The PHQ-8 is an eight-item, self-administered scale based on DSM-IV diagnostic criteria for major depression, identical to the PHQ-9 but without the suicide item. Each item is scored on a four-point scale with responses ranging from 0 (not at all) to 3 (nearly every day), assessing depression symptom frequency over the past two weeks. Total scores range from 0-24. A PHQ-8 score of 10 or more has been found to have 88% sensitivity and 88% specificity for diagnosis of major depression based on clinical interview. This measure captures depression as a healing outcome related to symptom reduction.
Generalized Anxiety Disorder-7 (GAD-7) | Baseline and 1-month follow-up (approximately 6-8 weeks after baseline)
  The GAD-7 is a 7-item self-report questionnaire for screening and measuring the severity of generalized anxiety disorder. Response options are identical to the PHQ-8, with items scored from 0 (not at all) to 3 (nearly every day), assessing anxiety symptom frequency over the past two weeks. Total scores range from 0 to 21, with scores of ≥5, ≥10, and ≥15 representing mild, moderate, and severe anxiety symptom levels, respectively. This measure captures anxiety as a healing outcome related to symptom reduction.
Trauma Recovery Actions Checklist (TRAC) | Baseline and 1-month follow-up (approximately 6-8 weeks after baseline)
  The TRAC is a 35-item checklist of recovery actions that participants are currently using, want to use, or do not want to use. The checklist provides a comprehensive assessment of various recovery strategies and actions. Subscales include: building positive emotions, sharing and connecting with others, reflecting and creating healing spaces, establishing security, and futuring (planning for the future). This measure captures the range of recovery actions participants are taking or considering to support their healing journey.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Sinko, PhD, MSHP, RN, Principal Investigator — Temple University
Locations (1):
- Women in Transition, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers due to the highly sensitive and potentially identifying nature of data collected from survivors of interpersonal violence. The study involves qualitative interviews, photographs, and detailed personal trauma histories that, even when de-identified, could pose risks to participant privacy and safety if shared. Protecting participant confidentiality is paramount given the vulnerable nature of this population and the potential for harm if participants were re-identified. However, aggregate data and de-identified findings will be disseminated through peer-reviewed publications, conference presentations, and reports to community partners as outlined in the study's dissemination plan.

REFERENCES:
- [Background] Sinko L, Saint Arnault D. Photo-experiencing and reflective listening: A trauma-informed photo-elicitation method to explore day-to-day health experiences. Public Health Nurs. 2021 Jul;38(4):661-670. doi: 10.1111/phn.12904. Epub 2021 Apr 4. PMID 33813744